CLINICAL TRIAL: NCT01639924
Title: Evaluation of Patients With Gastrointestinal Disease
Brief Title: Evaluation of People With Gastrointestinal Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120154; 12-DK-0154
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Gastrointestinal Diseases
Keywords: Upper GI Disease; Small Bowel Disease; Digestive Disease; Gastrointestinal Disease; Lower GI Disease; Natural History
MeSH Terms: conditions — Gastrointestinal Diseases; Digestive System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Cohort: Patients with known or suspected gastrointestinal disease

SUMMARY:
Background:

- Gastrointestinal diseases and disorders affect the throat, stomach, and intestines. There are many different kinds of these diseases. Clinical trials are being developed to study new ways to treat them. People who are interested in clinical trials need to be screened before they can take part in the studies. Researchers want to evaluate people with different stomach and intestine disorders to see if they are eligible for clinical trials.

Objectives:

- To study people who have gastrointestinal disorders and see if they are eligible for clinical trials.

Eligibility:

- Individuals at least 18 years of age who have or may have a gastrointestinal disorder.

Design:

* Participants will be screened with a physical exam and medical history. Blood, urine, and stool samples will be collected. Imaging studies such as x-rays and ultrasound will check to see if the disorder has affected other organs.
* Participants may have tests as needed depending on their disorder. These tests include the following:
* Colonoscopy and endoscopy of the large intestine, esophagus, and stomach.
* Stomach acid analysis to look at stomach pH levels.
* Wireless capsule endoscopy to take pictures of the small intestine.
* Hydrogen breath testing to study issues like bloating, diarrhea, and constipation.
* Sitz Marker Study to see how fast stool moves through the colon.
* Participants may donate extra blood, urine, or stool samples for study. They may also donate stomach contents or tissue from the gut.
* Treatment will not be provided as part of this study. However, participants may be admitted to other clinical trials.

DETAILED DESCRIPTION:
Patients with suspected or established acute or chronic gastrointestinal diseases are evaluated and treated in this protocol and will be screened for entry into other research protocols. This protocol serves several purposes: 1) allows for detailed inquiry into the gastrointestinal disorders of these patients and the status of other organ systems that would determine their ability to safely enroll in active Digestive Diseases Branch (DDB) research protocols; 2) allows investigators to offer clinical diagnostic testing, procedures, and treatment to patients if clinically indicated to facilitate their participation in clinical trials; 3) allows outpatient evaluation and treatment of patients with a variety of gastrointestinal diseases for the purposes of physician education in our accredited gastroenterology training program; and 4) After completion of the initial evaluation process, patients will either be offered a chance to participate in an active research protocol or, if no appropriate protocol is identified, patients may be seen long-term to follow the disease progression for potential future participation in DDB gastrointestinal studies. Recommendations for other treatment options outside of the NIH will be discussed with study patients and/or to their primary or referring physicians.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Known or suspected gastrointestinal disorders.
* Patients greater than or equal to 18 years of age capable of providing informed consent.
* Existence of a referring community physician who would be able to manage care outside of the NIH.

EXCLUSION CRITERIA:

* Significant medical illnesses that the investigators feel may interfere with potential evaluations.
* Any medical, psychiatric, or social conditions which, in the opinion of the investigators, would make participation in this protocol not in the best interest of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known or suspected gastrointestinal disease.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 2761 (Actual)
Dates: Start 2012-07-27 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Patients with gastrointestinal disease | until protocol closes
  screening protocol for gastrointestinal diseases.

SECONDARY OUTCOMES:
Allow outpatient evaluation and follow-up of patients with a variety of gastrointestinal diseases for the purposes of physician education in the NIDDK's accredited gastroenterology training program. | until protocol closes
  evaluation and follow-up of gastrointestinal diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Kumar, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2012-DK-0154.html